CLINICAL TRIAL: NCT04676932
Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory in Reducing Pain and Comfort on Women Undergoing Hysterosalpingography
Brief Title: Hysterosalpingography and Comfort Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sümeyye BAL (Other)
Responsible Party: Sponsor-Investigator, Sümeyye BAL, Lecturer, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020/41
Record Dates: First submitted 2020-11-30; First posted 2020-12-21 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Nursing Caries
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Type of intervention, testing the comfort and components of women undergoing Hysterosalpingography with Nursing Care Based on Kolcaba's Comfort Theory
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: participant women, care provider and Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing Care Based on Kolcaba's Comfort Theory (Experimental): In this study, nursing care based on Kolcaba's Comfort Theory will be applied to the intervention groups.
  Care will given when women after receiving the HSG attendance appointment. Care will terminated on the 15 minutes after the end of HSG undergoing.
  The time of the study 1-3 days for each women. Intervention Nursing Care Based on Kolcaba's Comfort Theory
  Interventions: Other: Nursing Care Based on Kolcaba's Comfort Theory
- Routine hospital schedule (No Intervention): The researcher sincerely answered all questions asked by the control group during the HSG period.

INTERVENTIONS:
Other: Nursing Care Based on Kolcaba's Comfort Theory — In this study, Nursing care based on Kolcaba's Comfort Theory will be applied for women undergoing HSG.
  Other Names: Comfort-oriented care , Mobile-assisted education and counselling, virtual reality glasses
  Arms: Nursing Care Based on Kolcaba's Comfort Theory

SUMMARY:
Hysterosalpingography (HSG) is the radiological evaluation of the uterine cavity and tubules by giving radiopaque material from the cervical canal to the uterine cavity. HSG is an invasive procedure and is often described by women as "uncomfortable, anxiety-inducing and painful", which indicates impaired comfort .Physical, emotional, sociocultural and environmental factors contribute to the formation of this condition. Comfort Theory is a nursing model that makes it easier for the caregivers to see their problems more systematically and to plan more easily. In the literature review, no studies have been found to determine the effect of Nursing Care Based on Kolcaba's Comfort Theory in Reducing Pain and Comfort on Women Undergoing Hysterosalpingography. It was aimed to determine the effect of Nursing Care Based on Kolcaba Comfort Theory on Pain and Comfort Level in Women Undergoing Hysterosalpingography Procedure.

Method. The universe of the research will form women applying for hysterosalpingography procedure in Turkey's northern province of the Health Research and Application Center between. The sample size to be taken from the universe was determined by power analysis based on the reference values of a similar study in the literature. According to the Power analysis, it was decided to include a total of 126 women, including 42 women, in each group (Control group, Intervention 1: Mobile-assisted education and counseling group, Intervention 2: Virtual reality glasses group). In this study, standard nursing care will be applied to the control group, and nursing care based on Kolcaba's Comfort Theory will be applied to the intervention groups.The data will be collected with the Visual Analog Scale(VAS) and General Comfort Questionnaire (GCQ)

DETAILED DESCRIPTION:
In this study, Nursing care based on Kolcaba's Comfort Theory will be applied for women undergoing HSG. Before the HSG , the women will be met at the appointment time and the women will be given care during the procedure.Up to 15 minutes after the procedure will be with women. There will be 2 intervention groups and one control group. In the first intervention group, virtual reality glasses will be applied during the procedure, Mobile-assisted education and consultancy will be provided in the 2nd intervention group. This mobile assisted education and consultancy starts 48 hours before HSG shooting.The hsg capture will continue until it ends. Hospital care standards will be applied to the control group, the third group.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in research
2. Being over 18 years old
3. To be at least a primary school graduate
4. To be able to read and write Turkish
5. Not having a diagnosed psychiatric disease
6. No mental deficiency and communication problems.
7. Drug sensitivity and lack of allergy
8. Regular menstrual cycle
9. Getting a diagnosis of primary infertility
10. Not having received infertility treatment before
11. Having a mobile phone capable of receiving and playing video messages

Exclusion Criteria:

1. Being illiterate
2. Being under the age of 18
3. Having a diagnosed psychiatric illness
4. Having mental deficiency and communication problems
5. Finding drug sensitivity and allergy
6. Diagnosing secondary infertility
7. Having an active genital infection
8. The absence of a mobile phone with the ability to receive and play video messages

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women Undergoing Hysterosalpingography
Enrollment: 126 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | 10 minutes
  After completing the HSG procedure, participants were asked to evaluate their pain in order to characterize pain intensity using the Visual Analog Scale (VAS). Patients indicated the maximum pain intensity experienced during the HSG by making a vertical line on the VAS.
  A standard ten-point visual analogue scale (VAS) of 0 to 10 was designed and used to assess the patients' perceptions of discomfort during the procedure. A high score on the scale indicated a high level of discomfort and a score of 0 denoted no discomfort at all. Patients indicate the degree of pain they feel between 0-10.
General Comfort Questionaire (GCQ) | 30 minutes
  The scale, which was developed by Katharine Kolcaba in 1992 in order to determine the comfort needs of individuals, to evaluate the nursing initiatives that can provide comfort and the increase in comfort, was adapted to Turkish society by Kuğuoğlu and Karabacak in 2004.The scale, which is a four-point Likert-type scale with 48 items, was created by guiding the taxonomic structure consisting of the theoretical components of comfort, including 3 levels and 4 dimensions. Level; While the dimension is evaluated as relief (16 items), relief (17 items) and overcoming the problems (15 items); It is evaluated in three parts: physical (12 items), psychospritual (13 items) and socio-cultural (10 items). Negative expressions in the scale are calculated by reverse coding during the evaluation phase. While the lowest total score that can be obtained from the scale is 48, the highest total score is 192.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krinsky R, Murillo I, Johnson J. A practical application of Katharine Kolcaba's comfort theory to cardiac patients. Appl Nurs Res. 2014 May;27(2):147-50. doi: 10.1016/j.apnr.2014.02.004. Epub 2014 Feb 14. PMID 24637106
- [Background] March A, McCormack D. Nursing theory-directed healthcare: modifying Kolcaba's comfort theory as an institution-wide approach. Holist Nurs Pract. 2009 Mar-Apr;23(2):75-80; quiz 81-2. doi: 10.1097/HNP.0b013e3181a1105b. PMID 19258847
- [Background] Koehn ML. Doğum ve doğum için alternatif ve tamamlayıcı tedaviler: Kolcaba'nın bütünsel konfor teorisinin bir uygulaması. Holist Hemşirelik Uygulaması. 2000 Ekim; 15 (1): 66-77. doi: 10.1097 / 00004650-200010000-00009. PMID: 12119621.
- [Background] Oliveira SM, Costa KNFM, Santos KFOD, Oliveira JDS, Pereira MA, Fernandes MDGM. Comfort needs as perceived by hospitalized elders: an analysis under the light of Kolcaba's theory. Rev Bras Enferm. 2020 Oct 19;73(suppl 3):e20190501. doi: 10.1590/0034-7167-2019-0501. eCollection 2020. English, Portuguese. PMID 33084827
- [Background] Wilson L, Kolcaba K. Practical application of comfort theory in the perianesthesia setting. J Perianesth Nurs. 2004 Jun;19(3):164-73; quiz 171-3. doi: 10.1016/j.jopan.2004.03.006. PMID 15195275
- [Derived] Bal S, Kulakac O. Effect of comfort theory-based nursing care on pain and comfort in women undergoing hysterosalpingography: a randomized controlled trial. Rev Assoc Med Bras (1992). 2023 Oct 30;69(12):e20230798. doi: 10.1590/1806-9282.20230798. eCollection 2023. PMID 37909532